CLINICAL TRIAL: NCT01470716
Title: A Phase II Study of Neo-adjuvant Erlotinib for Operable Stage IIB or IIIA Non-small Cell Lunc Cancer With Epidermal Growth Factor Receptor Activation Mutations
Brief Title: Neoadjuvant Erlotinib for Operable Stage II or IIIA NSCLC With EGFR Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Ji-youn Han, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-11-561
Record Dates: First submitted 2011-11-04; First posted 2011-11-11 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: NSCLC Stage II; NSCLC, Stage IIIA
Keywords: EGFR mutation; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study arm (Experimental): Neo-adjuvant Erlotinib treatment arm.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Neo-adjuvant Erlotinib treatment during maximum 8 weeks.
  Other Names: treatment arm

SUMMARY:
This study examines preoperative Erlotinib in patients with operable stage II and IIIA Non-small-cell lung cancer (NSCLC) harboring EGFR mutations.

DETAILED DESCRIPTION:
Lung cancer remains the most common cause of cancer-related death in the world. Non-small-cell lung cancer (NSCLC) is the most common type, and it accounts for 85% of cases. Unfortunately, the majority of patients with NSCLC have metastatic disease at diagnosis. However, even patients with resectable disease have poor survival. The need to improve survival rates in these patients prompted research exploring the role of systemic therapy in operable NSCLC. In the 1990s, several clinical trials of preoperative chemotherapy (also known as induction chemotherapy) followed by surgery or radiation in patients with locally advanced NSCLC showed improvements in survival. Erlotinib is an orally administered tyrosine kinase inhibitor of the epidermal growth factor receptor (EGFR). The presence of somatic mutations in the kinase domain of EGFR strongly correlates with increased responsiveness to EGFR tyrosine kinase inhibitors. Recently three randomized phase III trials showed that first-line use of EGFR-TKIs in patients with EGFR mutant NSCLC significantly improved response rate and progression-free survival (PFS) compared to platinum-based chemotherapy. These findings prompted this phase II trial of preoperative Erlotinib in patients with operable stage II and IIIA NSCLC harboring EGFR mutations.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed stage II & IIIA non-small cell lung cancer

  * EGFR exon 19 or 21 mutations
  * Age ≥ 18 years and ECOG performance 0~1
  * Has measurable lesion by RECIST 1.1
  * No previous chemotherapy or radiation therapy
  * Adequate organ function by following; ANC ≥1,500/uL, hemoglobin ≥9.0g/dL, platelet ≥100,000/uL, PaO2 ≥ 60 mmHg, Serum Cr < 1 x UNL or creatinine clearance > 60 ml/min, Serum bilirubin < 1 x UNL, AST (SGOT) and ALT (SGPT) < 2.5 x UNL, alkaline phosphatase < 5 x UNL
  * Written informed consent form

Exclusion Criteria:

* Previous chemotherapy or radiation therapy
* Previous history of malignancy within 5 years from study entry except treated non-melanomatous skin cancer or uterine cervical cancer in situ
* Known allergic history of erlotinib
* Interstitial lung disease or fibrosis on chest radiogram
* Active infection, uncontrolled systemic disease (cardiopulmonary insufficiency, fatal arrhythmias, hepatitis)
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free survival | every 8 week
  Progression free survival will be calculated from the date of study treatment start to the first objective documentation of progressive disease or to the date of death, whichever occurs first.

SECONDARY OUTCOMES:
Response rate | every 4 weeks
  The response rate will be determined by the number of patients with complete and partial responses according to RECIST criteria 1.1
Overall Survival Rate | every 3months, until death
  Survival time will be calculated from the date of study treatment start to the date of death.( or date last seen )
Toxicity profile | Every 4 weeks
  Safety will be evaluated by the frequency, severity, and relationship of adverse event graded by NCI Common Toxicity Criteria version 4.0 that occur during the treatment and follow up periods.

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Youn Han, M.D. PhD., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea